CLINICAL TRIAL: NCT02501993
Title: Serology Screening Test for the Detection of Nasopharyngeal Carcinoma in Zhongshan City
Brief Title: Nasopharyngeal Carcinoma Screening in Zhongshan City
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Mingfang Ji, Principal Investigator, Zhongshan People's Hospital, Guangdong, China
Other Study IDs: NPC-PRO-002
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening cohort: All participants will be tested for anti-EBV antibody by using serum samples. Participants are stratified into those having high, moderate and low antibody levels, those having moderate antibody levels are invited to retest annually in the following 3 years and those found to have high antibody levels on these occasions are referred to centers for diagnostic workup for NPC.

SUMMARY:
The primary objective is to determine the early diagnosis rate and mortality rate of the Nasopharyngeal Carcinoma (NPC) in the study population.

The secondary objective is to determine the incidence of NPC in the study population.

DETAILED DESCRIPTION:
The research is to evaluate the effect of NPC screening, also as an extended study of Screening for Nasopharyngeal Carcinoma in High Risk Populations (NCT00941538).

The program was conducted in Xiaolan and Minzhong towns of Zhongshan city in 2012.

All participants will be tested for anti-EBV antibody by using serum samples. Participants are stratified into those having high, moderate and low antibody levels, those having moderate antibody levels are invited to retest annually in the following 3 years and those found to have high antibody levels on these occasions are referred to centers for diagnostic workup for NPC.

ELIGIBILITY:
Inclusion Criteria:

* Subject residents in Zhongshan city
* Subject is 30 to 59 years of age inclusive
* Subject has no medical record of nasopharyngeal carcinoma
* ECOG 0-2
* Subject has psychical condition and well consciousness
* Subject is able to comprehend, sign, and date the written informed consent document to participate in the study.

Exclusion Criteria:

* Subject has heavy cardiovascular, liver or kidney disease
* Subject has medical record of nasopharyngeal carcinoma
* Subject who is not residing in Zhongshan City

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Zhongshan City
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The early detection rate (stage I and II) of Nasopharyngeal Carcinoma | 10 years
The mortality rate of Nasopharyngeal Carcinoma | 10 years

SECONDARY OUTCOMES:
The incidence of Nasopharyngeal Carcinoma | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mingfang Ji, MD, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan People's Hospital, Zhongshan, Guangdong, China